CLINICAL TRIAL: NCT07003633
Title: Preoperative Analgesia: The Effect of the Pericapsular Nerve Group (PENG) Block Administered Preoperatively in Patients With Hip Fractures on Preoperative Analgesic Efficacy, Early Postoperative Discharge, Mortality, and Morbidity.
Brief Title: Preoperative Analgesia: The Effectiveness of the PENG Block in Patients With Hip Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Alim Miniksar, MD, Anesthesiology and Reanimation Resident, M.D., Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-43012747-050.04-463726-205
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hip Fracture Surgeries
Keywords: Analgesia; PENG block; Hip Fracture
MeSH Terms: conditions — Agnosia; Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be randomized to their rescpective groups with closed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PENG (Experimental): Group PENG will involve the patients who will be performed PENG block 24 hours before surgery.
  Interventions: Procedure: PENG block with 0.25% bupivacaine guided by ultrasound.
- Group Control (No Intervention): Group Control will involve the patients who will not be performed PENG block preoperatively.

INTERVENTIONS:
Procedure: PENG block with 0.25% bupivacaine guided by ultrasound. — PENG (Pericapsular nerve block) is a peripheral nerve block which is performed for patients with hip fractures aimed to prevent preoperative and postoperative pain. It is performed under sterile conditions under ultrasound guideance.
  Arms: Group PENG

SUMMARY:
The aim is to provide effective preoperative analgesia in patients undergoing surgical procedures due to hip fractures by administering a pericapsular nerve group (PENG) block under ultrasound guidance. This approach seeks to increase patient satisfaction, reduce analgesic requirements, enable earlier discharge, and decrease morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip farcture surgery

Exclusion Criteria:

* Chronic analgesics consumption
* Patients contraindicated for neuraxial anesthesia
* Alcohol and drug addiction
* Allergies to local anesthetics and opioids
* Patients who refuses to participate in the study

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative Pain Scores and Opioid Consumption | 24 hours preoperatively
  Preoperative pain of patients will be assessed with NRS (Numeric Raitng Scale) which ranges from 0 (no pain) to 10 (the most severe pain imaginable).

SECONDARY OUTCOMES:
Discharge Time | From surgery to discharge up to 30 days
Postoperative Mortality and Morbidity | 30 days after surgery
  Postoperative complications such as infections, embolism, chronic pain and survival status
Opioid Consumption | 24 hours preoperatively
  Opioid consumption will be assessed with patient controlled analgesia (PCA) device which measures analgesic drug consumption. Fentanyl consumption unit will be micrograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Universtiy Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided